CLINICAL TRIAL: NCT05237167
Title: Time to Diagnosis of Glenohumeral Joint Dislocations in the Emergency Department- Traditional Radiography Versus Point-of-care Ultrasound
Brief Title: Time to Diagnosis of Glenohumeral Joint Dislocations in the ED- Traditional Radiography vs. POC Ultrasound
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was ultimately found to be too difficult to enroll patients and have an adequate control.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0790-21-FB
Record Dates: First submitted 2022-01-17; First posted 2022-02-11 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Glenohumeral Dislocation
Keywords: glenohumeral dislocation; POC Ultrasound; Plain radiograph
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Intervention Model Description: Prospective randomized diagnostic comparison study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Experimental): After randomization, these subjects will undergo diagnostic point-of-care ultrasound
  Interventions: Procedure: Shoulder reduction
- Radiograph (Active Comparator): After randomization, these subjects will undergo diagnostic plain radiograph
  Interventions: Procedure: Shoulder reduction

INTERVENTIONS:
Procedure: Shoulder reduction — This is standard of care and only measure as a time component outcome in the study

SUMMARY:
This is study to compare the time to diagnosis of glenohumeral joint dislocation using two imaging methods, traditional x-ray and point-of-care ultrasound. Participants who present at the emergency department complaining of shoulder injury and who are suspected of having a possible glenohumeral shoulder dislocation will be eligible for the study. A reduction of the joint will be performed if imaging findings so indicate. All participants will receive a post-reduction x-ray and be referred to appropriate follow-up care.

DETAILED DESCRIPTION:
This is a prospective comparison study evaluating the time to diagnosis of glenohumeral joint dislocation using two imaging modalities, traditional x-ray and point-of-care ultrasound. Eligible participants will include those who present to the emergency department with complaints of shoulder injury who are suspected by triage nursing of having a possible glenohumeral shoulder dislocation. Eligible participants will be consented by participating physicians and randomized into ultrasound or x-ray groups. If indicated based on the imaging findings, a reduction of the joint will be performed. All patients will receive a post-reduction x-ray and be referred to appropriate follow-up care based on the findings of their evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (19 and older in state of Nebraska) who present to the emergency department with shoulder pain/injury and potential shoulder dislocation

Exclusion Criteria:

* Injury sustained in major traumatic event (trauma activation), unable to consent, in extremis, less then 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis of glenohumeral joint dislocations | 0 to 60 minutes
  Comparison between point-of-care ultrasound and plain radiograph in time to diagnosis of glenohumeral joint dislocations who present to the emergency department

SECONDARY OUTCOMES:
Time to reduction of dislocation joint | 1 to 6 hours
  Time from presentation in Emergency Department to treatment (reduction of joint dislocation)
Emergency Department Length of Stay | 1 to 12 hours
  Total time in Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Bradford C Huff, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No
There is no currently plan to share IPD with other researchers.

REFERENCES:
- [Background] Secko MA, Reardon L, Gottlieb M, Morley EJ, Lohse MR, Thode HC Jr, Singer AJ. Musculoskeletal Ultrasonography to Diagnose Dislocated Shoulders: A Prospective Cohort. Ann Emerg Med. 2020 Aug;76(2):119-128. doi: 10.1016/j.annemergmed.2020.01.008. Epub 2020 Feb 25. PMID 32111508
- [Background] Kanji A, Atkinson P, Fraser J, Lewis D, Benjamin S. Delays to initial reduction attempt are associated with higher failure rates in anterior shoulder dislocation: a retrospective analysis of factors affecting reduction failure. Emerg Med J. 2016 Feb;33(2):130-3. doi: 10.1136/emermed-2015-204746. Epub 2015 Jun 25. PMID 26113487
- [Background] Gottlieb M, Russell F. Diagnostic Accuracy of Ultrasound for Identifying Shoulder Dislocations and Reductions: A Systematic Review of the Literature. West J Emerg Med. 2017 Aug;18(5):937-942. doi: 10.5811/westjem.2017.5.34432. Epub 2017 Jul 10. PMID 28874947
- [Background] Abbasi S, Molaie H, Hafezimoghadam P, Zare MA, Abbasi M, Rezai M, Farsi D. Diagnostic accuracy of ultrasonographic examination in the management of shoulder dislocation in the emergency department. Ann Emerg Med. 2013 Aug;62(2):170-5. doi: 10.1016/j.annemergmed.2013.01.022. Epub 2013 Mar 13. PMID 23489654
- [Background] Lahham S, Becker B, Chiem A, Joseph LM, Anderson CL, Wilson SP, Subeh M, Trinh A, Viquez E, Fox JC. Pilot Study to Determine Accuracy of Posterior Approach Ultrasound for Shoulder Dislocation by Novice Sonographers. West J Emerg Med. 2016 May;17(3):377-82. doi: 10.5811/westjem.2016.2.29290. Epub 2016 Apr 26. PMID 27330675
- [Background] Akyol C, Gungor F, Akyol AJ, Kesapli M, Guven R, Cengiz U, Toksul HI, Eken C. Point-of-care ultrasonography for the management of shoulder dislocation in ED. Am J Emerg Med. 2016 May;34(5):866-70. doi: 10.1016/j.ajem.2016.02.006. Epub 2016 Feb 16. PMID 26935225